CLINICAL TRIAL: NCT03871595
Title: Relative Bioavailability of BI 894416 as Tablet Formulation Following a High-fat, High-calorie Breakfast Compared to Administration in the Fasting State in Healthy Male Subjects (an Open-label, Randomised, Single-dose, Two-period, Two-sequence Crossover Study)
Brief Title: A Study in Healthy Men to Test Whether Food Affects the Amount of BI 894416 in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1371-0021; 2018-004313-41 (EudraCT Number)
Record Dates: First submitted 2019-03-11; First posted 2019-03-12 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2022-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BI 894416 30 mg fed (T) (Experimental): 3 tablets with 10 milligram (mg) of BI 894416 (total: 30 mg) were administered as one single oral dose with 240 milliliter (mL) of water after a high-fat, high-calorie meal (fed conditions) as test treatment (T).
  Interventions: Drug: BI 894416
- BI 894416 30 mg fast (R) (Experimental): 3 tablets with 10 milligram (mg) of BI 894416 (total: 30 mg) were administered as one single oral dose with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (fasted conditions) as reference treatment (R).
  Interventions: Drug: BI 894416

INTERVENTIONS:
Drug: BI 894416 — 3 tablets with 10 milligram (mg) of BI 894416 (total: 30 mg) were administered as one single oral dose with 240 milliliter (mL) of water.

SUMMARY:
Investigate the relative bioavailability of BI 894416 as tablet formulation following a high-fat, high calorie breakfast (Test, T) compared with administration in the fasting state (Reference, R)

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 50 years (inclusive)
* BMI of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with GCP and local legislation

Exclusion Criteria:

* Any finding in the medical examination (including Blood Pressure (BP), Pulse Rate (PR) or Electrocardiogram (ECG) and including the neurological examination) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause QT/QTc interval prolongation)
* Intake of an investigational drug in another clinical trial within 60 days of planned administration of investigational drug in the current trial, or concurrent participation in another clinical trial in which investigational drug is administered
* Smoker (unless the subject quit smoking for at least 3 months prior to first planned administration of trial medication)
* Alcohol abuse (consumption of more than 24 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days of planned administration of trial medication or intended blood donation during the trial
* Intention to perform excessive physical activities within one week prior to the administration of trial medication or during the trial
* Inability to comply with the dietary regimen of the trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant Electrocardiogram (ECG) finding at screening
* A history of additional risk factors for Torsade de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because the subject is not considered able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study

In addition, the following trial-specific exclusion criteria apply:

* History of relevant neurological disorder affecting the peripheral or central nervous system (this includes, but is not limited to: stroke, epilepsy, inflammatory or atrophic diseases affecting the nervous system, cluster headache or any cancer of the nervous system). Febrile seizures in childhood or adolescence, recovered carpal tunnel syndrome, recovered uncomplicated meningitis, recovered herpes zoster, tension headache, occasional benign tics (e.g. due to stress) or minor par- or dysesthesia (e.g. as a side effect of prior blood withdrawal) do not constitute a history of relevant neurological disorder.
* History of immunological disease except allergy not relevant to the trial (such as mild hay fever or dust mite allergy) and except asthma in childhood or adolescence
* History of cancer (other than successfully treated basal cell carcinoma)
* Male subjects with WOCBP partner who are unwilling to use male contraception (condom or sexual abstinence) from time point of first administration of trial medication until 30 days after the last administration of trial medication
* Further exclusion criteria apply

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2019-04-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A randomised, open-label, two-sequence crossover, single-dose, two-period trial in healthy male subjects to compare the test treatment (T) to the reference treatment (R). The treatments were 2 single oral doses of BI 894416 , administered under fasted (R) and fed (T) conditions and separated by a wash-out period of at least 5 days.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- 30 mg of BI 894416 Fasted - 30 mg of BI 894416 Fed: 3 tablets with 10 milligram (mg) of BI 894416 (total: 30 mg) were administered as one single oral dose with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (fasted conditions) as reference treatment (R) followed by a wash-out period of at least 5 days followed by 3 tablets with 10 mg of BI 894416 (total: 30 mg) administered as a single oral dose with 240 mL of water 30 minutes after a high-fat, high-calorie meal (fed conditions) as test treatment (T).
- 30 mg of BI 894416 Fed - 30 mg of BI 894416 Fasted: 3 tablets with 10 milligram (mg) of BI 894416 (total: 30 mg) were administered as one single oral dose with 240 milliliter (mL) of water after a high-fat, high-calorie meal (fed conditions) as test treatment (T) followed by a wash-out period of at least 5 days followed by 3 tablets with 10 mg of BI 894416 (total: 30 mg) administered as a single oral dose with 240 mL of water 30 minutes after an overnight fast of at least 10 hours (fasted conditions) as reference treatment (R).
Period: Treatment Period 1 (P1) + Wash-out
Arm/Group | 30 mg of BI 894416 Fasted - 30 mg of BI 894416 Fed | 30 mg of BI 894416 Fed - 30 mg of BI 894416 Fasted
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: Treatment Period 2 (P2)
Arm/Group | 30 mg of BI 894416 Fasted - 30 mg of BI 894416 Fed | 30 mg of BI 894416 Fed - 30 mg of BI 894416 Fasted
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The treated set included all subjects who received at least one dose of trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | 30 mg of BI 894416 Fasted - 30 mg of BI 894416 Fed | 30 mg of BI 894416 Fed - 30 mg of BI 894416 Fasted | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (5.1) | 41.4 (8.7) | 36.4 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 7 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of BI 894416 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of BI 894416 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz).
  Time points of pharmacokinetic (PK) blood samples are given as planned time relative to start of drug administration.
Time Frame: Within 3 hours before and then 15 minutes (min), 30 min, 45 min, and 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 34 and 48 hours after drug administration.
Population: The pharmacokinetic set included all subjects who received at least one dose of trial medication and provided at least one PK endpoint that was defined as primary and that was not excluded due to relevant protocol deviations or due to PK non-evaluability.
Measure: Geometric Mean (Standard Error); unit: nanomole (nmol) * hour (h) / liter (L)
Arm/Group | BI 894416 30 mg Fed (T) | BI 894416 30 mg Fast (R)
Number analyzed (Participants) | 14 | 14
nanomole (nmol) * hour (h) / liter (L) | 4436.69 (NA) — Standard Error is Geometric standard error (gSE) = 1.05. | 4458.63 (NA) — Standard Error is Geometric standard error (gSE) = 1.05.
Statistical Analysis 1: Comparison: BI 894416 30 mg Fed (T) vs BI 894416 30 mg Fast (R); Exploratory trial, no formal hypotheses were tested. Analysis of Variance (ANOVA) model on the logarithmic scale was used which included effects accounting for sources of variation: 'sequence' (fixed effect), 'subjects within sequences' (random effect), 'period' (fixed effect) and 'treatment' (fixed effect); Test type: Other — Relative bioavailability; Adjusted Geometric Mean Ratio T/R [%] = 99.51, 90% CI 2-sided [95.36 to 103.83], Standard Deviation 6.3 — The Adjusted Geometric Mean is adjusted by treatment. The standard deviation is actually the intraindividual geometric Coefficient of Variation [%]

2. Primary Outcome: Maximum Measured Concentration of BI 894416 in Plasma (Cmax)
Description: Maximum measured concentration of BI 894416 in plasma (Cmax). Time points of pharmacokinetic (PK) blood samples are given as planned time relative to start of drug administration.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: nanomole (nmol) / liter (L)
Arm/Group | BI 894416 30 mg Fed (T) | BI 894416 30 mg Fast (R)
Number analyzed (Participants) | 14 | 14
nanomole (nmol) / liter (L) | 492.90 (NA) — Standard Error is Geometric standard error (gSE) = 1.06. | 703.05 (NA) — Standard Error is Geometric standard error (gSE) = 1.06.
Statistical Analysis 1: Comparison: BI 894416 30 mg Fed (T) vs BI 894416 30 mg Fast (R); [analysis description as in outcome 1, analysis 1]; Test type: Other — Relative bioavailability; Adjusted Geometric Mean Ratio T/R [%] = 70.11, 90% CI 2-sided [62.67 to 78.44], Standard Deviation 16.8 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Area Under the Concentration-time Curve of BI 894416 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞ )
Description: Area under the concentration-time curve of BI 894416 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞ ).
  Time points of pharmacokinetic (PK) blood samples are given as planned time relative to start of drug administration.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: nanomole (nmol) * hour (h) / liter (L)
Arm/Group | BI 894416 30 mg Fed (T) | BI 894416 30 mg Fast (R)
Number analyzed (Participants) | 14 | 14
nanomole (nmol) * hour (h) / liter (L) | 4463.26 (NA) — Standard Error is Geometric standard error (gSE) = 1.05 | 4472.94 (NA) — Standard Error is Geometric standard error (gSE) = 1.05
Statistical Analysis 1: Comparison: BI 894416 30 mg Fed (T) vs BI 894416 30 mg Fast (R); [analysis description as in outcome 1, analysis 1]; Test type: Other — Relative bioavailability; Adjusted Geometric Mean Ratio T/R [%] = 99.78, 90% CI 2-sided [95.64 to 104.11], Standard Deviation 6.3 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From drug administration until the next drug administration or end of trial, up to 15 days.
Description: The treated set included all subjects who received at least one dose of trial medication.
Arm/Group | BI 894416 30 mg Fed (T) | BI 894416 30 mg Fast (R)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 1/14 | 3/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 894416 30 mg Fed (T) (N=14) | BI 894416 30 mg Fast (R) (N=14)
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/95/NCT03871595/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-03): https://cdn.clinicaltrials.gov/large-docs/95/NCT03871595/SAP_001.pdf